CLINICAL TRIAL: NCT04831788
Title: Pneumococcal Nasopharyngeal and Oropharyngeal Carriage in Adults Older Than 50 Years of Age in Outpatient Health Care Facility in Novi Sad
Brief Title: Pneumococcal Nasopharyngeal and Oropharyngeal Carriage in Adults
Status: Completed | Type: Observational
Sponsor: University of Novi Sad (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Vladimir Petrovic, Professor, University of Novi Sad
Other Study IDs: 01-1093/2
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-01

CONDITIONS: Preference, Patient
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Adults older than 50 years of age, residing in the city of Novi Sad, Serbia and providing oropharyngeal and nasopharyngeal swab specimen upon signing informed consent

SUMMARY:
This is the first baseline pilot-study that will evaluate the NP and OP colonization with the underline of pneumococcal serotype distribution among adults older than 50 years of age in Serbia and Southeastern Europe. Results of this project will serve as additional evidence in order to increase coverage among adults and elderly

DETAILED DESCRIPTION:
Research center(s):

The research will be carried out by the:

1. Institute of Public Health of Vojvodina

   * Centre for Disease Control and Prevention and the Centre for Microbiology
2. Health Care Centre of Novi Sad

   * Department of General Medicine.

Sample processing To confirm the NP and OP carriage, sampling will include NP and OP swabs. Swabs will be collected by the general practitioners in the Health Care Centre of Novi Sad and will transport, within 24h of collection, to the Centre for Microbiology of Institute of Public Health of Vojvodina, Novi Sad. The sterile cotton-tipped wire swabs will be inserted into the anterior nares, gently rubbed on the NP swab wall and immediately placed in transport medium (Copan Venturi Transystem, Brescia, Italy).

Laboratory procedure Within the laboratory NP swabs will be analyzed by 200 μl of swab-inoculated STGG media will be transferred to 5.0 ml Todd Hewitt broth containing 0,5% yeast extract (THY) and 1 ml of rabbit serum and incubated at 35-37 °C for six hours. Cultured broth will be plated on sheep blood agar and incubated in 5% CO2 at 35-37 °C. After 18-24 hours of incubation, plates will be examined for the appearance of alpha-haemolytic colonies resembling streptococci. Positive samples will be cultured, and optochin disc and bile solubility test will be performed.

Molecular serotyping

DNA Extraction To obtain DNA extracts for PCR reactions, an overnight growth of blood agar plate will be suspended in in 300 μl of 0.85% NaCl, heated to 70 °C for 15 min, spinned for 2 min and supernatant will be removed. Pellet will be suspended in 50 μl TE buffer with an addition of 10 μl mutanolysin and 8 μl of hyaluronidase, kept at 37°C for 30 min (to overnight), heated for 10 min at 100°C and spinned for 4 min. No more than 2,5 μl of supernatant will be used as DNA template. Extracts will be stored at -20°C until PCR testing (9).

Identification of S. pneumoniae Identification of S. pneumoniae will be achieved by amplifying the lytA gene using primers and probes recommended by CDC and Quanta Biosciences PerfeCTa1 qPCR ToughMix1, Low RoxTM (Quanta Biosciences, Beverly, USA) (10). LytA positive samples will be further analyzed for serotype identification.

Serotype identification Conventional multiplex PCR assays will be performed as a series of multiplex reactions, using CDC recommended schemes and primers for pneumococcal serotype deduction and 2X PCR Buffer - QIAGEN Multiplex PCR Kit (Qiagen, Hilden, Germany). The PCR products will be analyzed on 2% NuSieve agarose gels (Cambrex Bio Science, Inc., Rockland, ME), stained with ethidium bromide. Gel images will be recorded BioDocAnalyze system (Analytik Jena, Jena, Germany).

Real Time PCR will be performed optionally in case of any difficulties with conventional PCR. IT will be performed, as a series of 21 monoplex assays encompassing 21 serotypes using CDC recommended schemes based on geographic prevalence of serotypes. The assays are multiplexed in a sequential triplex format (three targets/serotypes in one reaction), each detecting targets on FAM, Rox (or Cy5) and Hex channels. Reactions will be performed on ABI 7500 Instruments (Thermo Fisher Scientific, Waltham, USA), using specific primers and probes and Invitrogen-Platinum Quantitive PCR SuperMix (Thermo Fisher Scientific, Waltham, USA).

Susceptibility testing Susceptibility of Spn isolates to Optochin, Oxacilin, Norfloxacin, Erytromycin, Clindamycin, Tetracycline and Trimetroprim-sulfometoxazole will be determined by the Diffusion method according to the European Committee on Antimicrobial Susceptibility Testing (EUCAST, www.eucast.org).

This baseline assessment is taking into consideration to present descriptive only current results, but they are not separately taken into account for comparative analysis.

The results of laboratory testing, conducted for each patient, will forwarded to elected physicians who indicated sampling of patient material.

Study procedures Adults will be recruited during their health examination at Health Care Centre of Novi Sad by their elected physician.

After providing a verbal and written explanation of the research aim (Appendix 1), informed consent (Appendix 2) will be obtained from subjects before enrolment. Personal and confidential information obtained from participants will be removed, except for demographic information, including date of sampling, age, gender, data on previous upper respiratory tract infection, number of children (siblings) aged 0-10 years residing in the household of participants with pneumococcal and influenza immunization history (because influenza immunization may prevent pneumococcal superinfections), smoking habits of participants and their household members and the information about home residence (Survey Questionnaire- Appendix 3).

Samples will be provided as one NP swab per study subject. Every participant will be assigned only once.

Confirmed case is every laboratory tested participant in which, after testing (PCR or ELISA), a positive result is obtained.

Statistical Analysis and Sample Size Justification Collection of the data Characteristics of all respondents acquired by questionnaire from Novi Sad, the test results of laboratory testing of samples of participants and the final characterization of Spn serotypes will be entered in specially designed database. Personal information of participants will be removed.

Investigator of the research along with statistician will analyze the collected data.

Sample size justification In accordance with the sample size calculation for a study estimating a population prevalence (11), between 350 and 500 samples are planned to be collected. If more than 500 will be eligible they will all be included. We presume to detect pneumococci in up to 10% PCR-positive to Spn. Total number of adults older than 50 years of age is around 120,000, and therefore we expect to collect the sample up to 0.4% of the total targeted population.

Expected results After carefully implementation of the research, we expected that Spn carriage among adults older than 50 years of age will be present in less than 10% of the total population. In addition, we presume that Spn serotypes covered by PPV or PCV will represent more than 60% and 50% of the serotypes in overall distribution among tested subjects.

Statistical Methods We will examine associations between risk factors and NP and OP carriage of pneumococci in participants aged older than 50 years. The following factors will be examined as possible risk factors in covered population: age, gender, data on previous upper respiratory tract infection, number of children (siblings) aged 0-10 years residing in the household of participants with pneumococcal and influenza immunization history, smoking habits of participants and their household members and the information about home residence. These factors will be analyzed by univariate and multivariate analyses (if appropriate). Also, the prevalence of NP and OP carriage as the proportion of participants whose nasopharyngeal cultures were positive for Spn and corresponding 95% confidence intervals will be estimated. All descriptive analyses will be performed using the SPSS Statistics software Version 21.0 (IBM Corp., Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 50 years of age visiting the Health Care Centre with or without signs of upper respiratory tract infection during the study period

Exclusion Criteria:

* Living outside of Novi Sad, use of oral antibiotics in the two weeks prior to taking the swab and presence of a confirmed immunodeficiency (hematological malignancies, inherited immunodeficiency, HIV, post-splenectomy status, cancer chemotherapy).

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target group of the research will be all adults who will visit their elected physicians in the Health Care Centre of Novi Sad (outpatient care facility). Only adults older than 50 years of age from Novi Sad with 341,624 (2011 Census) inhabitants will be recruited in this research.
  All patients older than 50 years of age will be interviewed by physicians at the admission. Nasopharyngeal and oropharyngeal swabs will be obtained and transported to the Institute of Public Health for the laboratory analyses.
Sampling Method: Non-Probability Sample
Enrollment: 521 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2022-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biljana Bozin, Ph.D, Study Director — University of Novi Sad, Medical Facultz
Locations (1):
- Health Care Centre Novi Sad, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: nasopharyngeal and oropharyngeal swab
Groups:
- Pneumococcal Nasopharyngeal and Oropharyngeal Carriage: Adults older than 50 years of age, residing in the city of Novi Sad, Serbia and providing oropharyngeal and nasopharyngeal swab specimen upon signing informed consent
Period: Overall Study
Arm/Group | Pneumococcal Nasopharyngeal and Oropharyngeal Carriage
Started | 521; 1042 nasopharyngeal and oropharyngeal swab
Completed | 521; 1042 nasopharyngeal and oropharyngeal swab
Not Completed | 0; 0 nasopharyngeal and oropharyngeal swab

BASELINE CHARACTERISTICS:
Population: Each participant provided one nasopharyngeal and one oropharyngeal swab
Arm/Group | Pneumococcal Nasopharyngeal and Oropharyngeal Carriage
Number analyzed (Participants) | 521
Age, Continuous [Median (Full Range); unit: years] — Median age of participants who were eligible . Youngest was 50 and oldest 93 years of age.
  years | 71 [50 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 324
  Male | 197
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 521
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Serbia | 521
Number of Participants [Number; unit: participants] — Number of people who provided samples. Each provided one nasopharyngeal and one oropharyngeal swab
  participants | 521

OUTCOME MEASURES:

1. Primary Outcome: Prevalence
Description: Prevalence will be measured as a number of participants with positive isolates divided with overall number of participants analyzed and multiplied by a hundred to determine a percentage of positives
Time Frame: 90 days
Population: Prevalence was measured as a percentage of participants with Spn positive isolates
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumococcal Nasopharyngeal and Oropharyngeal Carriage
Number analyzed (Participants) | 521
Participants | 16

2. Secondary Outcome: Number of Participants With Spn Serotypes
Description: Serotype on NP and OP carriage with pneumococcal serotypes among adults older than 50 years of age in the city of Novi Sad according to specific clinical indications set for the PPV or PCV
Time Frame: 150 days
Population: participants with Spn positive isolates
Measure: Count of Participants; unit: Participants
Groups:
- Pneumococcal Nasopharyngeal and Oropharyngeal Carriage: Subset of participants with Spn serotype isolated (16) among overall number of participants (521)
Arm/Group | Pneumococcal Nasopharyngeal and Oropharyngeal Carriage
Number analyzed (Participants) | 16
Participants
  Non Typeable serotypes | 10
  Typeable serotypes | 6

ADVERSE EVENTS:
Time Frame: No adverse events were followed
Description: No adverse events were followed because this was not interventional study. No drugs or vaccines were investigated.
  This was observational study and mortality was not measure of outcome.
Arm/Group | Adults
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT04831788/Prot_SAP_ICF_000.pdf